CLINICAL TRIAL: NCT01458106
Title: An Open-Label, Multicenter Evaluation of Safety, Pharmacokinetics, and Efficacy of Recombinant Coagulation Factor VIII Fc Fusion Protein, BIIB031, in the Prevention and Treatment of Bleeding Episodes in Pediatric Subjects With Hemophilia A
Brief Title: Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of Recombinant Coagulation Factor VIII Fc Fusion Protein (rFVIIIFc) in Previously Treated Pediatric Subjects With Hemophilia A
Acronym: Kids ALONG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bioverativ Therapeutics Inc. (Industry)
Collaborators: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8HA02PED; 2011-003073-28
Record Dates: First submitted 2011-10-20; First posted 2011-10-24 (Estimated); Results first posted 2014-12-12 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2018-08

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — factor VIII-Fc fusion protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All participants (Experimental): PK subgroup: After a Washout Period of ≥72 hours, at the Baseline Visit (28±7 days prior to Day 1), participants receive a single IV injection of prestudy FVIII over 5 (±2) minutes at a dose of 50 IU/kg, rounded up to the nearest 250 IU increment, for a PK assessment. Following a second Washout Period of ≥72 hours, participants receive a single IV injection of rFVIIIFc over 5 (±2) minutes at a dose of 50 IU/kg for PK assessment. The first prophylactic dose of rFVIIIFc is administered at a starting dose of 25 IU/kg IV injection on Day 1 and 50 IU/kg on Day 4. Dose increases to a maximum of 80 IU/kg, and frequency of administration to a minimum interval of once every 2 days, are allowed as indicated.
  Non-PK subgroup: On Day 1, a first prophylactic dose of rFVIIIFc of 25 IU/kg IV injection is given, followed by a dose of 50 IU/kg on Day 4. Dose increases to a maximum of 80 IU/kg, and frequency of administration to a minimum interval of once every 2 days, are allowed as indicated.
  Interventions: Drug: BIIB031 (rFVIIIFc); Drug: FVIII (PK subgroup only)

INTERVENTIONS:
Drug: BIIB031 (rFVIIIFc) — Vials of rFVIIIFc were combined as needed, based on the actual labeled potency to achieve the participant's calculated dose. Partial vial use was allowed, in order to achieve the calculated dose.
  Other Names: ELOCTATE; efmoroctocog alfa; antihemophilic factor (recombinant), Fc fusion protein; recombinant coagulation factor VIII Fc fusion protein
Drug: FVIII (PK subgroup only) — Baseline prestudy FVIII dosing in participants who enter the PK subgroup. Vials of prestudy FVIII were combined as needed, based on the nominal labeled potency (e.g., 250 IU, 500 IU, and 1000 IU), to achieve the participant's calculated dose.

SUMMARY:
The primary objective of the study is to evaluate the safety of Recombinant Coagulation Factor VIII Fc Fusion Protein (rFVIIIFc) in previously treated pediatric subjects with hemophilia A. Secondary objectives of this study in this study population are as follows: to evaluate the efficacy of rFVIIIFc for prevention and treatment of bleeding episodes; to evaluate and assess the pharmacokinetics (PK) of rFVIIIFc; and to evaluate rFVIIIFc consumption for prevention and treatment of bleeding episodes.

DETAILED DESCRIPTION:
Previously treated pediatric participants will be treated with a prophylactic regimen of rFVIIIFc. PK analysis of pre-study factor VIII (FVIII) and rFVIIIFc will be performed in a sub-group of the study participants prior to commencement of prophylactic treatment. After these PK results are available, remaining participants have the option of proceeding directly to prophylactic treatment. After completing the end of study assessments, eligible participants would be able to continue treatment in Study 8HA01EXT.

ELIGIBILITY:
Key Inclusion Criteria:

* Severe hemophilia A defined as <1 IU/dL (<1%) endogenous FVIII
* Male <12 years of age and weight ≥13 kg
* History of at least 50 documented prior exposure days to FVIII
* No current, or history of, inhibitor development to FVIII

Key Exclusion Criteria:

* Other coagulation disorders in addition to Hemophilia A
* History of anaphylaxis associated with any FVIII or IV immunoglobulin administration

NOTE: Other protocol-defined Inclusion/Exclusion criteria may apply.

Max Age: 11 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 71 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Bioverativ Therapeutics Inc.
Locations (23):
- United States (12):
  - Research Site, Los Angeles, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, Aurora, Colorado
  - Research Site, Chicago, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, St Louis, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Pittsburgh, Pennsylvania
- Australia (2):
  - Research Site, Brisbane, Queensland
  - Research Site, Melbourne, Victoria
- Research Site, Hong Kong, Hong Kong
- Research Site, Dublin, Ireland
- Research Site, Groningen, Netherlands
- Research Site, Lublin, Poland
- Research Site, Johannesburg, South Africa
- United Kingdom (4):
  - Research Site, Cambridge, Cambridgshire
  - Research Site, Basingstoke, Hampshire
  - Research Site, Glasgow
  - Research Site, London

REFERENCES:
- [Derived] Raheja P, Kragh N, Bystricka L, Eriksson D, Aroui K, Mezghani M, Barbier S, Linari S. Long-term efmoroctocog alfa prophylaxis improves perceived pain, mental, and physical health in patients with hemophilia A: post hoc analysis of phase III trials using patient-reported outcomes. Ther Adv Hematol. 2024 Jul 30;15:20406207241257917. doi: 10.1177/20406207241257917. eCollection 2024. PMID 39091324
- [Derived] Katragadda S, Neelakantan S, Diao L, Wong N. Population Pharmacokinetic Analysis of Recombinant Factor VIII Fc Fusion Protein in Subjects With Severe Hemophilia A: Expanded to Include Pediatric Subjects. J Clin Pharmacol. 2021 Jul;61(7):889-900. doi: 10.1002/jcph.1854. Epub 2021 Apr 14. PMID 33719084
- [Derived] Young G, Mahlangu J, Kulkarni R, Nolan B, Liesner R, Pasi J, Barnes C, Neelakantan S, Gambino G, Cristiano LM, Pierce GF, Allen G. Recombinant factor VIII Fc fusion protein for the prevention and treatment of bleeding in children with severe hemophilia A. J Thromb Haemost. 2015 Jun;13(6):967-77. doi: 10.1111/jth.12911. Epub 2015 Apr 23. PMID 25912075

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants < 6 Years Old: Pharmacokinetic (PK) subgroup: After a Washout Period of ≥72 hrs, at the Baseline Visit (28±7 days prior to Day 1), participants receive a single IV injection of prestudy FVIII over 5±2 minutes at a dose of 50 IU/kg, rounded up to the nearest 250 IU increment, for PK assessment. Following a second Washout Period of ≥72 hrs, participants receive a single IV injection of rFVIIIFc over 5±2 mins at a dose of 50 IU/kg for PK assessment. The first prophylactic dose of rFVIIIFc is administered at a starting dose of 25 IU/kg IV injection on Day 1 and 50 IU/kg on Day 4. Dose increases to a maximum of 80 IU/kg, and frequency of administration to a minimum interval of once every 2 days, are allowed as indicated.
  Non-PK subgroup: On Day 1, a first prophylactic dose of rFVIIIFc of 25 IU/kg IV injection is given, followed by a dose of 50 IU/kg on Day 4. Dose increases to a maximum of 80 IU/kg, and frequency of administration to a minimum interval of once every 2 days, are allowed as indicated.
- Participants 6 to < 12 Years Old: PK subgroup: After a Washout Period of ≥72 hours, at the Baseline Visit (28±7 days prior to Day 1), participants receive a single IV injection of prestudy FVIII over 5 (±2) minutes at a dose of 50 IU/kg, rounded up to the nearest 250 IU increment, for a PK assessment. Following a second Washout Period of ≥72 hours, participants receive a single IV injection of rFVIIIFc over 5 (±2) minutes at a dose of 50 IU/kg for PK assessment. The first prophylactic dose of rFVIIIFc is administered at a starting dose of 25 IU/kg IV injection on Day 1 and 50 IU/kg on Day 4. Dose increases to a maximum of 80 IU/kg, and frequency of administration to a minimum interval of once every 2 days, are allowed as indicated.
  Non-PK subgroup: On Day 1, a first prophylactic dose of rFVIIIFc of 25 IU/kg IV injection is given, followed by a dose of 50 IU/kg on Day 4. Dose increases to a maximum of 80 IU/kg, and frequency of administration to a minimum interval of once every 2 days, are allowed as indicated.
Period: Overall Study
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Started | 36 | 35
PK Subgroup | 25 | 35
Non-PK Subgroup | 11 | 0
Completed | 33 | 34
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Pre-rFVIIIFc Adverse Event | 1 | 0
Not completed — Withdrawn Per Protocol | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Participants < 6 Years Old; Participants 6 to < 12 Years Old: PK subgroup: After a Washout Period of ≥72 hours, at the Baseline Visit (28±7 days prior to Day 1), participants receive a single IV injection of prestudy FVIII over 5 (±2) minutes at a dose of 50 IU/kg, rounded up to the nearest 250 IU increment, for a PK assessment. Following a second Washout Period of ≥72 hours, participants receive a single IV injection of rFVIIIFc over 5 (±2) minutes at a dose of 50 IU/kg for PK assessment. The first prophylactic dose of rFVIIIFc is administered at a starting dose of 25 IU/kg IV injection on Day 1 and 50 IU/kg on Day 4. Dose increases to a maximum of 80 IU/kg, and frequency of administration to a minimum interval of once every 2 days, are allowed as indicated.
  Non-PK subgroup: On Day 1, a first prophylactic dose of rFVIIIFc of 25 IU/kg IV injection is given, followed by a dose of 50 IU/kg on Day 4. Dose increases to a maximum of 80 IU/kg, and frequency of administration to a minimum interval of once every 2 days, are allowed as indicated.
- Total: Total of all reporting groups
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old | Total
Number analyzed (Participants) | 36 | 35 | 71
Age, Continuous [Median (Full Range); unit: years] | 4.0 [1 to 5] | 8.0 [6 to 11] | 5.0 [1 to 11]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 36 | 35 | 71

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of FVIII Inhibitor Development
Description: An inhibitor test result ≥0.6 Bethesda units (BU)/mL, confirmed on 2 separate samples drawn 2 to 4 weeks apart, was considered positive. Both tests were to be performed by the central laboratory using the Nijmegen-modified Bethesda Assay. Incidences were summarized for any positive inhibitor for participants with ≥50 EDs to rFVIIIFc. In addition, the incidence for all participants, regardless of their EDs to rFVIIIFc, was also summarized. An exact 95% CI for the proportion of participants with a confirmed inhibitor was calculated using the Clopper-Pearson exact method for a binomial proportion.
Time Frame: Up to Week 26 +/- 7 days, or up to 50 exposure days (EDs) if reached prior to Week 26
Population: Safety Analysis Set: participants who received at least 1 dose of prestudy FVIII, or at least 1 dose of rFVIIIFc; n=number of participants with given number of exposure days who had a valid inhibitor test.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old | All Arms: Total
Number analyzed (Participants) | 36 | 35 | 71
percentage of participants
  Participants with ≥50 EDs; n=27, 34, 61 | 0 [0 to 12.77] | 0 [0 to 10.28] | 0 [0 to 5.87]
  All participants; n=36, 35, 71 | 0 [0 to 9.74] | 0 [0 to 10.00] | 0 [0 to 5.06]

2. Secondary Outcome: Annualized Bleeding Rate
Description: Annualized bleeding rate = (number of bleeding episodes during the efficacy period / total number of days during the efficacy period)*365.25. The efficacy period begins with the first prophylactic dose of rFVIIIFc and ends with the last dose (for prophylaxis or a bleed). Surgery/rehabilitation periods and PK evaluation periods are not included in the efficacy period. A bleeding episode started from the first sign of a bleed and ended no more than 72 hours after the last treatment for the bleed, within which any symptoms of bleeding at the same location or injections less than or equal to 72 hours apart were considered the same bleeding episode. Any injection to treat the bleeding episode taken more than 72 hours after the preceding one was considered the first injection to treat a new bleeding episode at the same location. Any bleeding at a different location was considered a separate bleeding episode, regardless of time from last injection.
Time Frame: Up to Week 26 +/- 7 days (efficacy period as defined in description)
Population: Full Analysis Set: participants who received at least 1 dose of rFVIIIFc; based on the number of participants whose efficacy period was of at least 1 day in duration.
Measure: Median (Inter-Quartile Range); unit: bleeding episodes per participant per yr
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 35 | 34
bleeding episodes per participant per yr | 0.00 [0.00 to 3.96] | 2.01 [0.00 to 4.04]

3. Secondary Outcome: Annualized Joint Bleeding Rate (Spontaneous)
Description: Annualized bleeding rate for spontaneous joint bleed=(number of bleeding episodes meeting those criteria during the efficacy period/total number of days during the efficacy period)*365.25. The efficacy period begins with the first prophylactic dose of rFVIIIFc and ends with the last dose (for prophylaxis or a bleed). Surgery/rehabilitation periods and PK evaluation periods are not included in the efficacy period. A bleeding episode started from the first sign of a bleed and ended no more than 72 hours after the last treatment for the bleed, within which any symptoms of bleeding at the same location or injections less than or equal to 72 hours apart were considered the same bleeding episode. Any injection to treat the bleeding episode taken more than 72 hours after the preceding one was considered the first injection to treat a new bleeding episode at the same location. Any bleeding at a different location was considered a separate bleeding episode, regardless of time from last inject
Time Frame: Up to Week 26 +/- 7 days (efficacy period as defined in description)
Population: Full Analysis Set: participants who received at least 1 dose of rFVIIIFc; based on the number of participants whose efficacy period is of at least 1 day in duration.
Measure: Median (Inter-Quartile Range); unit: bleeding episodes per participant per yr
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 35 | 34
bleeding episodes per participant per yr | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]

4. Secondary Outcome: Participant Assessment of Response to Injections to Treat a Bleeding Episode
Description: Participant's assessment (provided by the caregiver) of the response to the first rFVIIIFc injection for each bleeding episode. Percentages were based on the number of first injections for which a response was provided, using the following 4-point scale: excellent=abrupt pain relief and/or improvement in signs of bleeding within approximately 8 hours after the initial injection; good=definite pain relief and/or improvement in signs of bleeding within approximately 8 hours after a single injection, but possibly requiring more than one injection after 24 to 48 hours for complete resolution; moderate=probable or slight beneficial effect within approximately 8 hours after the initial injection and requiring more than one injection; no response=no improvement, or condition worsened, within approximately 8 hours after the initial injection.
Time Frame: Up to Week 26 +/- 7 days
Population: Full Analysis Set: participants who received at least 1 dose of rFVIIIFc and had a bleeding episode; participants with a non-evaluable bleed are counted in the number of participants analyzed, but not the percentages.
Measure: Number; unit: percent of 1st injections w/ a response
Units Other Than Participants: Injections
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 17 | 20
Number analyzed (Injections) | 35 | 46
percent of 1st injections w/ a response
  Excellent or Good | 91.4 | 93.5
  Excellent | 65.7 | 47.8
  Good | 25.7 | 45.7
  Moderate | 8.6 | 2.2
  No Response | 0 | 4.3

5. Secondary Outcome: Physician's Global Assessment of the Participant's Response to His rFVIIIFc Regimen
Description: Investigators assessed each participant's response to his rFVIIIFc regimen using a 4-point scale: excellent=bleeding episodes responded to ≤ the usual number of injections or ≤ the usual dose of rFVIIIFc or the rate of breakthrough bleeding during prophylaxis was ≤ that usually observed; effective=most bleeding episodes responded to the same number of injections and dose, but some required more injections or higher doses, or there was a minor increase in the rate of breakthrough bleeding; partially effective=bleeding episodes most often required more injections and/or higher doses than expected, or adequate breakthrough bleeding prevention during prophylaxis required more frequent injections and/or higher doses; ineffective=routine failure to control hemostasis, or hemostatic control required additional agents. Percentages are based on the total number of responses; multiple responses per participant are counted.
Time Frame: Up to Week 26 +/- 7 days
Population: Full Analysis Set: participants who received at least 1 dose of rFVIIIFc; based on the number of responses.
Measure: Number; unit: percentage of responses
Units Other Than Participants: Responses
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 35 | 34
Number analyzed (Responses) | 141 | 165
percentage of responses
  Excellent | 96.5 | 89.7
  Effective | 3.5 | 9.1
  Partially Effective | 0 | 1.2
  Ineffective | 0 | 0

6. Secondary Outcome: Annualized rFVIIIFc Consumption Per Participant
Description: Consumption is calculated for the efficacy period. The efficacy period begins with the first prophylactic dose of rFVIIIFc and ends with the last dose (for prophylaxis or a bleed). Surgery/rehabilitation periods and PK evaluation periods are not included in the efficacy period. Annualized consumption = (total IU/kg of study treatment received during the efficacy period / total number of days during the efficacy period)*365.25. Consumption was calculated overall for all participants and for the last 3 months (91 days) on study, counted backwards from the end of the efficacy period, for participants with at least 24 weeks on study.
Time Frame: Up to Week 26 +/- 7 days (efficacy period as defined in description)
Population: Full Analysis Set: participants who received at least 1 dose of rFVIIIFc. 'Overall' n=participants in the Full Analysis Set with evaluable data in the efficacy period; 'Last 3 Months on Study' n=participants in the Full Analysis Set with evaluable data and ≥ 24 weeks on study.
Measure: Mean (Standard Deviation); unit: IU/kg rFVIIIFc per participant per year
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 35 | 34
IU/kg rFVIIIFc per participant per year
  Overall (n=35, 34) | 5331.8 (1106.68) | 4973.5 (976.06)
  Last 3 months on study (n=26, 33) | 5562.1 (1474.42) | 5092.6 (1013.01)

7. Secondary Outcome: Number of Days From Last Treatment Injection to a Spontaneous Bleeding Episode
Description: The number of days from the last prophylaxis injection to the onset of a new spontaneous bleeding episode, analyzed across all evaluable bleeding episodes per participant and per episode, based on the efficacy period. Evaluable bleeding episodes are those for which both a date and time are available for both the onset of the bleeding episode and the previous prophylactic injection. The efficacy period begins with the first prophylactic dose of rFVIIIFc and ends with the last dose (for prophylaxis or a bleed). Surgery/rehabilitation periods and PK evaluation periods are not included in the efficacy period. For 'Per participant' values, the number of days from the last prophylactic injection to a spontaneous bleeding episode is averaged across all evaluable spontaneous bleeding episodes per participant.
Time Frame: Up to Week 26 +/- 7 days (efficacy period as defined in description)
Population: Full Analysis Set: participants who received at least 1 dose of rFVIIIFc; number of participants and number of episodes were determined for participants with at least 1 evaluable spontaneous bleeding episode.
Measure: Median (Inter-Quartile Range); unit: days
Units Other Than Participants: Evaluable Spontaneous Bleeding Episodes
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 8 | 7
Number analyzed (Evaluable Spontaneous Bleeding Episodes) | 17 | 19
days
  Per Participant | 2.17 [1.51 to 2.84] | 2.55 [1.58 to 3.04]
  Per Spontaneous Bleeding Episode | 2.16 [1.35 to 2.87] | 2.77 [1.58 to 3.29]

8. Secondary Outcome: Number of Injections Required for Resolution of a Bleeding Episode
Description: The number of injections required to resolve a bleeding episode per participant and per episode, based on the efficacy period. The efficacy period begins with the first prophylactic dose of rFVIIIFc and ends with the last dose (for prophylaxis or a bleed). Surgery/rehabilitation periods and PK evaluation periods are not included in the efficacy period. All injections given from the initial sign of a bleed, until the last date/time within the bleed window are counted. The resolution of a bleed is defined as no sign of bleeding following injection for the bleed. For 'Per participant' values, the number of injections required to resolve each bleed is averaged across all bleeding episodes per participant.
Time Frame: Up to Week 26 +/- 7 days (efficacy period as defined in description)
Population: Full Analysis Set: participants who received at least 1 dose of rFVIIIFc; number of participants and number of episodes were determined for participants with at least 1 evaluable bleeding episode.
Measure: Median (Inter-Quartile Range); unit: injections
Units Other Than Participants: Bleeding Episodes
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 17 | 20
Number analyzed (Bleeding Episodes) | 38 | 48
injections
  Per Participant | 1.0 [1.0 to 1.2] | 1.0 [1.0 to 1.2]
  Per Bleeding Episode | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]

9. Secondary Outcome: Total Dose Required for Resolution of a Bleeding Episode
Description: The total dose required to resolve a bleeding episode per participant and per episode, based on the efficacy period. The efficacy period begins with the first prophylactic dose of rFVIIIFc and ends with the last dose (for prophylaxis or a bleed). Surgery/rehabilitation periods and PK evaluation periods are not included in the efficacy period. For 'Per bleeding episode' values, for each bleeding episode, the total dose is the sum of the doses (IU/kg) administered across all injections given to treat that bleeding episode. For 'Per participant' values, the total dose (IU/kg) used to resolve each bleed is averaged across all bleeding episodes per participant.
Time Frame: Up to Week 26 +/- 7 days (efficacy period as defined in description)
Population: Full Analysis Set: participants who received at least 1 dose of rFVIIIFc; number of participants and number of episodes were determined for participants who had complete information on the dose administered to treat a bleeding episode.
Measure: Median (Full Range); unit: IU/kg
Units Other Than Participants: Bleeding Episodes
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 17 | 20
Number analyzed (Bleeding Episodes) | 38 | 48
IU/kg
  Per Participant | 55.56 [22.6 to 150.7] | 51.35 [20.1 to 152.3]
  Per Bleeding Episode | 56.40 [13.9 to 200.0] | 53.49 [14.0 to 196.6]

10. Secondary Outcome: Maximum Plasma Activity (Cmax; One-stage Activated Partial Thromboplastin Time [aPTT] Clotting Assay)
Description: Maximum plasma activity during a dosing interval for participants in the PK subgroup. The values for Cmax were adjusted to the nominal dose of 50 IU/kg. The 95% confidence interval on the geometric mean is based on the t-statistic back-transformed from the log scale.
Time Frame: Baseline (28 ±7 days prior to Day 1) Prestudy FVIII Dosing: predose; 30 ±5 min, 3 hours ±30 min, 24 ±3 hours, 48 ±4 hours post-dose. Day 1 (rFVIIIFc Dosing): predose; 30 ±5 min, 3 hours ±30 min, 24 ±3 hours, 48 ±4 hours, 72 ±7 hours post-dose
Population: PK Analysis Set: All participants in the PK subgroup with adequate PK data, defined as complete and evaluable PK samples through 72 hours after rFVIIIFc dosing. Complete means the availability of the 72-hour sample and at least enough other samples to allow for all the PK parameters to be estimated.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/dL
Groups:
- Participants < 6 Years Old; Participants 6 to < 12 Years Old: PK subgroup: After a Washout Period of ≥72 hours, at the Baseline Visit (28±7 days prior to Day 1), participants receive a single IV injection of prestudy FVIII over 5 (±2) minutes at a dose of 50 IU/kg, rounded up to the nearest 250 IU increment, for a PK assessment. Following a second Washout Period of ≥72 hours, participants receive a single IV injection of rFVIIIFc over 5 (±2) minutes at a dose of 50 IU/kg for PK assessment. The first prophylactic dose of rFVIIIFc is administered at a starting dose of 25 IU/kg IV injection on Day 1 and 50 IU/kg on Day 4. Dose increases to a maximum of 80 IU/kg, and frequency of administration to a minimum interval of once every 2 days, are allowed as indicated.
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 23 | 31
IU/dL | 95.03 [89.23 to 101.21] | 114.94 [102.13 to 129.35]

11. Secondary Outcome: Maximum Plasma Activity (Cmax; Two-stage Chromogenic Assay)
Description: as for outcome 10
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: IU/dL
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 24 | 27
IU/dL | 94.11 [86.40 to 102.51] | 103.80 [95.68 to 112.60]

12. Secondary Outcome: Elimination Half Life (t1/2; One-stage aPTT Clotting Assay)
Description: Time required for the activity of the drug to reach half of its original value for participants in the PK subgroup. The 95% confidence interval on the geometric mean is based on the t-statistic back-transformed from the log scale.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 23 | 31
hours | 12.277 [10.988 to 13.718] | 13.451 [11.445 to 15.808]

13. Secondary Outcome: Elimination Half Life (t1/2; Two-stage Chromogenic Assay)
Description: as for outcome 12
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 24 | 27
hours | 14.268 [12.559 to 16.210] | 15.861 [13.814 to 18.210]

14. Secondary Outcome: Clearance (CL; One-stage aPTT Clotting Assay)
Description: Rate at which the body removes the drug, measured as the volume of the plasma cleared of drug per unit time per unit weight for participants in the PK subgroup. The 95% confidence interval on the geometric mean is based on the t-statistic back-transformed from the log scale.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: mL/h/kg
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 23 | 31
mL/h/kg | 3.4561 [3.0564 to 3.9080] | 2.6067 [2.2559 to 3.0119]

15. Secondary Outcome: Clearance (CL; Two-stage Chromogenic Assay)
Description: as for outcome 14
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: mL/h/kg
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 24 | 27
mL/h/kg | 3.8600 [3.4839 to 4.2767] | 3.0486 [2.6187 to 3.5491]

16. Secondary Outcome: Volume at Steady State (Vss; One-stage aPTT Clotting Assay)
Description: Volume of distribution at steady state for participants in the PK subgroup. The 95% confidence interval on the geometric mean is based on the t-statistic back-transformed from the log scale.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: mL/kg
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 23 | 31
mL/kg | 57.94 [54.13 to 62.01] | 49.51 [44.08 to 55.60]

17. Secondary Outcome: Volume at Steady State (Vss; Two-stage Chromogenic Assay)
Description: as for outcome 16
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: mL/kg
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 24 | 27
mL/kg | 66.48 [59.77 to 73.93] | 63.15 [56.26 to 70.87]

18. Secondary Outcome: Dose Normalized Area Under the Curve (DNAUC; One-stage aPTT Clotting Assay)
Description: Dose normalized area under the FVIII activity-time curve for participants in the PK subgroup. The 95% confidence interval on the geometric mean is based on the t-statistic back-transformed from the log scale.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: IU*h/dL per IU/kg
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 23 | 31
IU*h/dL per IU/kg | 28.93 [25.59 to 32.72] | 38.37 [33.20 to 44.35]

19. Secondary Outcome: Dose Normalized Area Under the Curve (DNAUC; Two-stage Chromogenic Assay)
Description: as for outcome 18
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: IU*h/dL per IU/kg
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 24 | 27
IU*h/dL per IU/kg | 25.90 [23.38 to 28.69] | 32.80 [28.18 to 38.19]

20. Secondary Outcome: Mean Residence Time (MRT; One-stage aPTT Clotting Assay)
Description: The average time that a drug molecule is present in the systemic circulation for participants in the PK subgroup. The 95% confidence interval on the geometric mean is based on the t-statistic back-transformed from the log scale.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 23 | 31
hours | 16.762 [15.106 to 18.599] | 18.999 [16.213 to 22.263]

21. Secondary Outcome: Mean Residence Time (MRT; Two-stage Chromogenic Assay)
Description: as for outcome 20
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 24 | 27
hours | 17.220 [15.407 to 19.246] | 20.708 [18.036 to 23.776]

22. Secondary Outcome: Incremental Recovery (IR; One-stage aPTT Clotting Assay)
Description: The rise in FVIII activity in IU/dL per unit dose administered in IU/kg for participants in the PK subgroup. The 95% confidence interval on the geometric mean is based on the t-statistic back-transformed from the log scale.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: IU/dL per IU/kg
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 23 | 31
IU/dL per IU/kg | 1.901 [1.785 to 2.024] | 2.299 [2.042 to 2.587]

23. Secondary Outcome: Incremental Recovery (IR; Two-stage Chromogenic Assay)
Description: as for outcome 22
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: IU/dL per IU/kg
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 24 | 27
IU/dL per IU/kg | 1.882 [1.728 to 2.050] | 2.076 [1.914 to 2.252]

24. Secondary Outcome: Time at Maximum Activity (Tmax; One-stage aPTT Clotting Assay)
Description: Time at which maximum activity (Cmax) is observed for participants in the PK subgroup. The 95% confidence interval on the geometric mean is based on the t-statistic back-transformed from the log scale.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 23 | 31
hours | 0.6987 [0.5256 to 0.9287] | 0.7257 [0.5685 to 0.9264]

25. Secondary Outcome: Time at Maximum Activity (Tmax; Two-stage Chromogenic Assay)
Description: as for outcome 24
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 24 | 27
hours | 0.7313 [0.5408 to 0.9889] | 0.6334 [0.5184 to 0.7741]

26. Secondary Outcome: Lambda Z (One-stage aPTT Clotting Assay)
Description: First order rate constant associated with the terminal portion of the curve (lambda z) for participants in the PK subgroup. The 95% confidence interval on the geometric mean is based on the t-statistic back-transformed from the log scale.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: 1/hours
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 23 | 31
1/hours | 0.05644 [0.05053 to 0.06304] | 0.05158 [0.04390 to 0.06061]

27. Secondary Outcome: Lambda Z (Two-stage Chromogenic Assay)
Description: as for outcome 26
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: 1/hours
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 24 | 27
1/hours | 0.04848 [0.04264 to 0.05511] | 0.04367 [0.03801 to 0.05018]

28. Secondary Outcome: Volume at Terminal Phase (Vz; One-stage aPTT Clotting Assay)
Description: Volume of distribution estimated from the terminal phase for participants in the PK subgroup. The 95% confidence interval on the geometric mean is based on the t-statistic back-transformed from the log scale.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: mL/kg
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 23 | 31
mL/kg | 61.22 [56.54 to 66.29] | 50.58 [44.54 to 57.43]

29. Secondary Outcome: Volume at Terminal Phase (Vz; Two-stage Chromogenic Assay)
Description: as for outcome 28
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: mL/kg
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 24 | 27
mL/kg | 79.48 [69.20 to 91.30] | 69.75 [62.98 to 77.25]

30. Secondary Outcome: Area Under the Curve to the Last Measurable Timepoint (AUClast; One-stage aPTT Clotting Assay)
Description: Dose-normalized area under the FVIII activity-time curve to the last measurable timepoint for participants in the PK subgroup. The 95% confidence interval on the geometric mean is based on the t-statistic back-transformed from the log scale.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: IU*h/dL
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 23 | 31
IU*h/dL | 1410.4 [1254.8 to 1585.2] | 1823.4 [1602.2 to 2075.0]

31. Secondary Outcome: Area Under the Curve to the Last Measurable Timepoint (AUClast; Two-stage Chromogenic Assay)
Description: as for outcome 30
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: IU*h/dL
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 24 | 27
IU*h/dL | 1250.1 [1133.2 to 1379.0] | 1540.4 [1346.5 to 1762.3]

32. Secondary Outcome: Area Under the Curve to Infinity (AUCinf; One-stage aPTT Clotting Assay)
Description: Dose normalized area under the FVIII activity-time curve to infinity for participants in the PK subgroup. The 95% confidence interval on the geometric mean is based on the t-statistic back-transformed from the log scale.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: IU*h/dL
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 23 | 31
IU*h/dL | 1446.5 [1279.2 to 1635.7] | 1918.5 [1660.0 to 2217.3]

33. Secondary Outcome: Area Under the Curve to Infinity (AUCinf; Two-stage Chromogenic Assay)
Description: as for outcome 32
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: IU*h/dL
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 24 | 27
IU*h/dL | 1294.7 [1168.7 to 1434.3] | 1640.0 [1408.7 to 1909.4]

34. Secondary Outcome: Percentage of AUCinf Extrapolated From the Last Data Point to Infinity (%AUCext; One-stage aPTT Clotting Assay)
Description: Percentage of AUCinf extrapolated from the last data point to infinity for participants in the PK subgroup. The 95% confidence interval on the geometric mean is based on the t-statistic back-transformed from the log scale.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: percentage of AUCinf
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 23 | 31
percentage of AUCinf | 1.8421 [1.3218 to 2.5673] | 2.7777 [1.9611 to 3.9344]

35. Secondary Outcome: Percentage of AUCinf Extrapolated From the Last Data Point to Infinity (%AUCext; Two-stage Chromogenic Assay)
Description: as for outcome 34
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: percentage of AUCinf
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 24 | 27
percentage of AUCinf | 2.7530 [2.1052 to 3.6001] | 3.9476 [2.8296 to 5.5074]

ADVERSE EVENTS:
Time Frame: Serious adverse events (AEs): from informed consent up to 21 days after last treatment visit (LTV); AEs: from Baseline (28 ± 7 days prior to Day 1) for PK Subgroup or from Day 1 (first dose of rFVIIIFc) for non-PK subgroup, up to 14 (+7) days after LTV.
Description: Length of rFVIIIFc dosing was up to 26 weeks ± 7 days. Serious and non-serious AEs that were treatment-emergent with respect to rFVIIIFc are presented for those participants who were treated with rFVIIIFc. Data are presented for the Full Analysis Set (participants who received at least 1 dose of rFVIIIFc).
Groups:
- Participants < 6 Years Old; Participants 6 to < 12 Years Old: PK subgroup: After a Washout Period of ≥ 72 hours, at the Baseline Visit (28 ± 7 days prior to Day 1), participants receive a single IV injection of prestudy FVIII over 5 (± 2) minutes at a dose of 50 IU/kg, rounded up to the nearest 250 IU increment, for a PK assessment. Following a second Washout Period of ≥ 72 hours, participants receive a single IV injection of rFVIIIFc over 5 (± 2) minutes at a dose of 50 IU/kg for PK assessment. The first prophylactic dose of rFVIIIFc is administered at a starting dose of 25 IU/kg IV injection on Day 1 and 50 IU/kg on Day 4. Dose increases to a maximum of 80 IU/kg, and frequency of administration to a minimum interval of once every 2 days, are allowed as indicated.
  Non-PK subgroup: On Day 1, a first prophylactic dose of rFVIIIFc of 25 IU/kg IV injection, followed by a dose of 50 IU/kg on Day 4. Dose increases to a maximum of 80 IU/kg, and frequency of administration to a minimum interval of once every 2 days, are allowed as indicated.
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Serious Adverse Events (participants affected / at risk) | 4/35 | 1/34
Other Adverse Events (participants affected / at risk) | 31/35 | 28/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants < 6 Years Old (N=35) | Participants 6 to < 12 Years Old (N=34)
Bacillus Infection (Infections and infestations) | 0 | 1
Croup Infectious (Infections and infestations) | 1 | 0
Escherichia Infection (Infections and infestations) | 0 | 1
Metapneumovirus Infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Head Injury (Injury, poisoning and procedural complications) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Participants < 6 Years Old (N=35) | Participants 6 to < 12 Years Old (N=34)
Ear Pain (Ear and labyrinth disorders) | 2 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 4
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 3 | 2
Fatigue (General disorders) | 1 | 3
Pyrexia (General disorders) | 1 | 2
Seasonal Allergy (Immune system disorders) | 2 | 2
Bronchitis (Infections and infestations) | 2 | 0
Conjunctivitis Infective (Infections and infestations) | 0 | 2
Ear Infection (Infections and infestations) | 2 | 2
Gastroenteritis (Infections and infestations) | 2 | 0
Nasopharyngitis (Infections and infestations) | 2 | 4
Otitis Media (Infections and infestations) | 2 | 0
Pharyngitis (Infections and infestations) | 2 | 2
Tonsillitis (Infections and infestations) | 2 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 7 | 2
Varicella (Infections and infestations) | 2 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 3 | 0
Face Injury (Injury, poisoning and procedural complications) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 3 | 2
Head Injury (Injury, poisoning and procedural complications) | 1 | 2
Limb Injury (Injury, poisoning and procedural complications) | 0 | 2
Lip Injury (Injury, poisoning and procedural complications) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Headache (Nervous system disorders) | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.